CLINICAL TRIAL: NCT05684978
Title: Efficacy and Safety of Perampanel in the Treatment of Refractory Status Epilepticus
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was not initiated.
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Maysaa Basha, Principle Investigator, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-22-05-4691
Record Dates: First submitted 2022-12-19; First posted 2023-01-13 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Refractory Status Epilepticus
Keywords: Status Epilepticus; Epilepticus; Epilepsy; Perampanel; Clinical trial for epilepsy; Epilepsy treatment; Seizure; seizure treatment; generalized tonic-clonic seizures; focal seizures; Refractory status epilepticus; (RSE); fycompa
MeSH Terms: conditions — Status Epilepticus; Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm prospective study (Experimental): * Adults patients equal or greater than 18 years
  * Patients in RSE that require IV anesthetic infusions. Note: RSE is defined as status epilepticus that fails to terminate after an adequate dose of benzodiazepines (1st line agents) and an AED (2nd line agent). Adequate doses have been defined in the screening (below).
  * Patients taking oral contraception who will be on the study long term should be informed about additional alternative methods of contraception.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — The purpose of this study is to determine the efficacy of Perampanel, an approved antiseizure medication, in the treatment of refractory status epilepticus (RSE), to identify determinants of outcomes, and establish safety.
  Other Names: Fycompa

SUMMARY:
This project is aiming to better understand the use of perampanel as an appropriate standard-of-care therapy for treatment refractory status epilepticus (RSE), to identify determinants of outcomes, and establish safety. The study will recruit 25 patients at WSU. The study will last for about 96 weeks and will involve a screening visit and two in clinic visits at 3 and 6 months. If the subjects give written informed consent and meet all eligibility criteria they will be clinically evaluated and will be given the study drug. This study will involve recording of patients medical history, drug history and epilepsy history. A physical exam and a and neurological exam will also be performed to study the heath status of the participant. Results and patient information will be stored in a database for analysis to find commonality among key factors that have been seen in past research.

DETAILED DESCRIPTION:
ILAE (International league against epilepsy) defines status epilepticus (SE) as generalized tonic-clonic seizures > 5 minutes or focal impaired awareness seizure > 15 min or recurrent seizures with alteration of consciousness in between seizures.

Refractory status epilepticus (RSE) is defined as failure to respond to first line benzodiazepines and one antiepileptic drug (AED). It often requires treatment with anesthetic drugs and continuous EEG monitoring for diagnosis and titration of medications. Status epilepticus (SE) is estimated to be refractory in about 30 % of cases, associated with increased morbidity and mortality and requires continuous EEG monitoring to guide treatment [1]. It is seen across all ages, and around 200,000 cases are seen in the United States annually resulting in significant morbidity and mortality [2]. Morbidity and mortality of SE and especially RSE is due to prolonged stay in the ICU and at times treatment from IV anesthetics including hemodynamic instability, and related infections of the ICU stays.

Standard of Care treatment of SE and RSE

Rapid termination of the SE is the primary goals of SE treatment with evidence indicating that if left untreated, SE becomes harder to terminate [3,4]. In a patient with SE, the first AED should be started at the onset concomitantly with the first line benzodiazepine or soon after. The agents of choice are typically those available in IV (intravenous) formulation with purpose of fast and safe administration in a seizing patient. These include phenytoin (PHT)/fosphenytoin, valproic acid (VPA), levetiracetam (LEV); lacosamide (LCM) with no clear evidence that one drug is superior [5,6]. Beyond the introduction of a second seizure medication, there is no unified consensus or clear evidence to guide treatment at that stage of RSE.

Other AED are used as add-on therapy in the treatment of SE when benzodiazepine (1st agent) and IV AED (2nd agent) fail. These have been demonstrated to be efficacious in different cohorts and case series and include but not limited to clobazam, topiramate, oxcarbazepine and eslicarbazepine [7].

Perampanel

Perampanel (PMP) has recently been shown to be efficacious in the treatment of variable subsets of SE including simple partial SE, refractory SE, and super-refractory SE [8, 9]. Efficacy of 75% was also demonstrated in a very difficult to treat subset of patient with nonconvulsive SE in post-anoxic patients. Systematic qualitative analysis of publications in use of PMP for status epilepticus revealed highly variable results in highly variable populations [10]. More homogeneous single-center outcomes are needed. In a multi-centered study looking at 52 patients receiving PMP for treatment of SE, PMP was the last drug added in 61.5 % of patients and a positive response attributed to PMP in 36.5% and PMP was well tolerated with minimal side effects and no discontinuation [11].

The mechanism of action unique to PMP may be key in its success in this disease state. Perampanel (PMP) is a selective noncompetitive AMPA receptor antagonist. Blockade of excitatory mechanisms become important in SE given that prolonged SE may result in postsynaptic internalization of GABA-A receptors and subsequent reduced efficacy of GABAergic drugs [12]. In addition, PMP is rapidly absorbed by the GI system and peak plasma concentrations are achieved as early as 0.5 hours (0.5-2.5hours) with 100% bioavailability; features which make the drug attractive even in its oral form in the treatment of SE.

Two studies (E2007-A001-024 and E2007-A001-023) in healthy recreational drug users evaluated safety and abuse potential of perampanel and submitted with PMP NDA (#202834) to the FDA. Data was established at 8mg, 24mg, and 36 mg in both studies (Table 1). Increasing the dose to 36 mg was not associated with significant safety or tolerability issues. [Somnolence and dizziness were the most common side effects. Hemodynamics (systolic blood pressure, diastolic blood pressure, and heart rate) were not impacted. Kidney and liver functions were also largely not impacted with the exception of a single-incident of liver enzyme elevation. In order to reach steady state, simulation data reveals that steady state is reached immediately with a 4-5:1 dosing (loading dose to maintenance dose) Thus, the established safety confirmed a 36 mg loading dose as safe and tolerable. Hence, the investigators have chosen this as the loading dose for our study. Given that this is not an FDA approved dosage or indication, the investigators have obtained FDA authorization as an investigational new drug (IND 157959) to conduct this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients equal or greater than 18 years
* Patients in RSE that require IV anesthetic infusions. Note: RSE is defined as status epilepticus that fails to terminate after an adequate dose of benzodiazepines (1st line agents) and an AED (2nd line agent). Adequate doses have been defined in the screening (below).
* Patients taking oral contraception who will be on the study long term should be informed about additional alternative methods of contraception.

Exclusion Criteria:

* Childbearing potential female who has a positive pregnancy test result or is otherwise known to be pregnant. Hypoglycemia or hyperglycemia induced seizures
* Mild, moderate or severe hepatic impairment
* Severe renal impairment or on hemodialysis
* History of psychiatric illness or suicidal behavior/ideation
* Previous or current use of PMP
* Known severe allergy to any AED
* Anoxic brain injury as etiology of status epilepticus
* Use caution in patients taking moderate and strong CYP3A4 Inducers (including carbamazepine, oxcarbazepine, and phenytoin)
* Patients on other forms of strong CYP3A4 (e.g. Rifampin, St John's Wart, etc).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes | Within 48 hours of stopping intravenous anesthetics
  Successful wean of IV anesthetics without recurrence of status epilepticus.
  a. Determined by absence of clinical and electrographic seizure activity.

SECONDARY OUTCOMES:
Secondary Outcomes | 3 months and 6 months
  1. Total duration of IV anesthetic infusion
  2. Number of AEDs used
  3. Number of intubation days
  4. ICU length of stay (LOS)
  5. Hospital LOS
  6. In hospital mortality
  7. Modified Rankin Scale (mRS) at discharge, 3 months and 6 months
  8. Extended Glasgow Outcome Scale (e-GOS) at discharge, 3 months and 6 months
  9. Discharge location
  10. Outpatient seizure control at 3 months and 6 months
2. Total duration of intravenous anesthetic infusion. | 90 Days
  a. Total length of IV anesthetic infusion usage in days
3. The number of antiseizure medications used. | 90 Days
  a. Determined by the number of antiseizure medications used during hospitalization.
3. Total duration of intubation | 90 days
  a. Total length of intubation in days
Total ICU and in-hospital length of stay | 90 days
  a. Total ICU and in-hospital length of stay in days
5. Mortality rate | ICU and hospital discharge
  Death rate
6. Functional impairment | Hospital discharge, 3 months, 6 months
  a. Percentage of patients that experience functional impairment as determined by modified Rankin Scale (mRS) during review of charts and/or general practitioner interview.
  Appendix 1. Modified Rankin Scale (MRS)
  Modified Ranking Scale Scale Symptom description 0 No symptoms
  1. No significant disability, despite symptoms; able to perform all usual duties and activities
  2. Slight disability; unable to perform all previous activities but able to look after own affairs without assistance
  3. Moderate disability; requires some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance
  5. Severe disability; bedridden, incontinent, and requires constant nursing care and attention
  6. Death
7. Favorable outcome | Hospital discharge, 3 months, 6 months
  A favorable outcome is defined by a Extended-Glasgow Outcome Scale (e-GOS).The Glasgow Outcome Scale (GOS) will be determined according to patients charts review and/or general practitioner interview conducted by an independent assessor.
  Appendix 2. Extended Glasgow Outcome Scale
  Extended Glasgow Outcome Scale (GOS-E) Category Description Death Dead Vegetative state (VS) Unable to obey commands Lower severe disability (LSD) Dependent on others for care Upper severe disability (USD) Independent at home Lower moderate disability (LMD) Independent at home and outside the home but with some physical or mental disability Upper moderate disability (UMD) Independent at home and outside the home but with some physical or mental disability, with less disruption than LMD Lower good recovery (LGR) Able to resume normal activities with some injury-related problems Upper good recovery (UGR) No injury-related problems.
8. Favorable discharge location | Hospital discharge
  Patients home or arranged living facility.
  1. Acute or subacute rehabilitation facility
  2. Nursing Facility
  3. Death unfavorable living location
Seizure Control | Determined by percentages of the patients that do not experience seizure recurrence
  Hospital discharge, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maysaa Basha, MD, Principal Investigator — Wayne State University; Wazim Mohamed, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data in accordance with clinical care will be collected through chart review. Long term Follow up Data collection will be prospectively collected in person and transferred into an Research Database.
  Once a subject is consented, the data to be collected will include the following variables:
  * Demographic data (age, sex, race/ethnicity)
  * Presumed etiology of SE
  * Neurological co-morbidities including prior history of epilepsy
  * Neurologic examination
  * Medical co-morbidities
  * Medication list
  * Social history including functional status, employment, and use of alcohol and drug use
  * EEG pattern of status epilepticus, duration of status epilepticus.
  * Neuroimaging reports
  * Treatment of SE details:
    * Medications and dosage
    * intubation and duration
    * complications and interventions (use of vasopressors and antibiotics)
  * Daily laboratory values including blood chemistry and hematology.